CLINICAL TRIAL: NCT03195205
Title: A Novel Approach Continuum to Identification to Elimination in HCV-Infected Individuals on Opioid Substitution Therapy and High-Risk Populations
Brief Title: Identification to Elimination in HCV-Infected Individuals
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: TruCare Internal Medicine & Infectious Disease (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Principal Investigator, Tuesdae Stainbrook, DO, MPH, Principal Investigator, TruCare Internal Medicine & Infectious Disease
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: GSI-2016-09-APR
Record Dates: First submitted 2017-05-31; First posted 2017-06-22 (Actual); Last update posted 2020-07-02 (Actual); Status verified 2020-07

CONDITIONS: Hepatitis C
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- High-Risk Patients (Other): OraQuick HCV screening for HCV-Infected Individuals on Opioid Substitution Therapy and High-Risk Populations
  Interventions: Diagnostic Test: OraQuick HCV Rapid Antibody Test

INTERVENTIONS:
Diagnostic Test: OraQuick HCV Rapid Antibody Test — HCV Screening

SUMMARY:
Approximately 3.5 - 5 million Americans are living with hepatitis C virus (HCV) in the United States. HCV significantly impacts rural Pennsylvania. It is estimated that 160,000 adults in Pennsylvania are living with hepatitis C. In 2010, Center for Rural Pennsylvania estimated that 27% of population of PA live in one of Pennsylvania's 48 rural counties. Under this estimate, there are over 43,000 individuals affected with chronic HCV living in rural Pennsylvania. Rural county residents often experience barriers to health care by having fewer primary care providers and limited specialty care physicians available to them to address their healthcare needs.

RQ1: Will the community based delivery system for Hepatitis C screenings see an increase in positivity rates?

HO1: There is no relationship between the community based delivery system with an increase in the Hepatitis C screening positivity rates.

HA1: There is a relationship between the community based delivery system with an increase in the Hepatitis C screening positivity rates.

DETAILED DESCRIPTION:
In rural Pennsylvania, transportation is considered a socioeconomic barrier and social detriment to personal health. Using an evidence-based model of population health by bringing the care into the high-risk population's community setting reduces the transportation and socioeconomic barriers of the most vulnerable at risk populations.

It is estimated that 35% to 65% of Opioid Substitution Treatment Patients (OST), are infected with HCV. Therefore, OPT programs that are already operating will be engaged and will be a primary focus for patient screening and recruitment for these services. In addition, high volume venues attracting high-risk populations will also be targeted to encourage HCV screening, education, and treatment.

Primary Objectives:

To screen Opioid Substitution Treatment Patients (OST), high-risk individual at Opioid Treatment Programs (OTP), and/or all high-risk populations in outlying sites (Anti-HCV prevalence)

To initiate HCV treatment of OST patients and other high-risk individuals at OTP facilities and/or high risk populations in outlying sites (linkage of care)

To maintain the successful HCV therapy and cure [Sustained Viral Response (SVR)] in OST patients and other high-risk individuals at OPT facility and/or high risk populations in outlying sites (retention)

To facilitate the use of a patient navigator and nursing case management staff to reduce barriers to initial screening and patient education

ELIGIBILITY:
Inclusion Criteria:

Subjects will be included in the study if the following criteria is met:

1. The subject must be an Opioid Substitution Treatment patient.
2. The subject must fall into another high-risk population for the HCV.

Exclusion Criteria:

Subjects may be excluded from the study if the subject falls into an exclusion category as identified as:

1. The subject cannot be or suspected of being pregnant
2. The subject cannot be under the age of 18 years.
3. No subjects requiring a legally authorized representative will be enrolled

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3051 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2020-04-20 (Actual); Study Completion 2020-04-20 (Actual)

PRIMARY OUTCOMES:
Positivity rates | 20 - 40 minutes
  The study will measure the percentage of patients screened for Hepatitis C who are reactive by detecting HCV antibodies.

SECONDARY OUTCOMES:
Linked to care | 1 - 3 months
  The study will measure the percentage of patients identified as reactive that follow up by linking to care.
Treatment | 8 - 24 weeks
  The study will measure the percentage of patients linked to care who complete treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Tuesdae R Stainbrook, DO, MPH, Principal Investigator — Trucare Internals Medicine & Infectious Disease
Locations (1):
- TruCare Internal Medicine & Infectious Diseases, DuBois, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided